CLINICAL TRIAL: NCT00612950
Title: Four Weeks of Near Normalisation of Blood Glucose Improves the Insulin Response to GLP-1 and GIP in Patients With Type 2 Diabetes
Brief Title: Beta-Cell Function After Near-Normalisation of Blood Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Patricia Verdugo Højberg/ MD, PHD, Kettegaard Alle 30, 2650 Hvidovre
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: KA 03005; KA 03005
Record Dates: First submitted 2008-01-16; First posted 2008-02-12 (Estimated); Last update posted 2008-02-12 (Estimated); Status verified 2008-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glucagon-Like Peptide 1; Incretins; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- GLP-1 (Experimental)
  Interventions: Drug: glucagon-like peptide-1,
- GIP (Experimental)
  Interventions: Drug: glucose dependent insulinotropic polypeptide
- saline (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: glucagon-like peptide-1, — GLP-1:continuous infusion of ½ pmol/kg/min for a total time of 120 minutes.
  Arms: GLP-1
Drug: glucose dependent insulinotropic polypeptide — continuous infusion of GIP (1½ pmol/kg/min) for 120 min.
  Arms: GIP
Drug: Saline — continuous infusion of Saline for 120 min
  Arms: saline

SUMMARY:
The incretin effect is attenuated in patients with type 2 diabetes mellitus partly due to impaired potentiation of beta-cell responsiveness to glucose by glucose dependent insulinotropic polypeptide and glucagon-like peptide-1 respectively. The aim of the present study was to investigate whether 4 weeks of near-normalization of blood glucose could improve the insulin responses to GIP and GLP-1 in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Type 2 diabetes diagnosed after 30 years of age
* BMI > 25

Exclusion Criteria:

* Severe complications to diabetes
* Abnormal liver and kidney function
* Haemoglobin below the lower limit
* Macroalbuminuria
* Systemic disease
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2006-10; Primary Completion 2007-02 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
2.phase insulin response measured as incremental area under the curve from 10-120 minutes | 2 hours

SECONDARY OUTCOMES:
2.phase insulin response measured as incremental area under the curve from 10-120 minutes, after 4 weeks of insulin treatment | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Patricia V Højberg, MD, PHD, Principal Investigator — University Hospital Hvidovre
Locations (1):
- Dept. of Endocrinology, Hvidovre Hospital, Copenhagen, Denmark

REFERENCES:
- [Derived] Hojberg PV, Vilsboll T, Rabol R, Knop FK, Bache M, Krarup T, Holst JJ, Madsbad S. Four weeks of near-normalisation of blood glucose improves the insulin response to glucagon-like peptide-1 and glucose-dependent insulinotropic polypeptide in patients with type 2 diabetes. Diabetologia. 2009 Feb;52(2):199-207. doi: 10.1007/s00125-008-1195-5. Epub 2008 Nov 27. PMID 19037628